CLINICAL TRIAL: NCT01673321
Title: Effect of Varied Protein Concentrations in Greek Yogurt on Glycemic Response, Satiety and Next Meal Food Intake in Healthy Young Men
Brief Title: Protein Concentrations in Yogurt and Satiety, Food Intake and Glycemia in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Dairy Farmers of Ontario (Other); Mondelēz International, Inc. (Industry)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 27226
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Healthy; Glucose Metabolism
Keywords: Yogurt; Milk; Protein; Food intake; Appetite; Glucose; Insulin
MeSH Terms: conditions — Insulin Resistance | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Non-fat Yogurt-Plain flavored (Experimental): Protein to carbohydrate ratio: 2.30
  Interventions: Other: Dietary intervention
- Skim milk (Experimental): Protein to carbohydrate ratio: 0.69
  Interventions: Other: Dietary intervention
- Non-fat Yogurt with honey-Plain flavored (Experimental): Protein to carbohydrate ratio: 1.24
  Interventions: Other: Dietary intervention
- Orange juice (Experimental): Protein to carbohydrate ratio: 0.07
  Interventions: Other: Dietary intervention
- Non-fat Yogurt-Strawberry flavored (Experimental): Protein to carbohydrate ratio: 0.79
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — All snacks (arms) were randomly given to subjects to be consumed within 5 minutes, after 4 hours of consuming a standard breakfast.

SUMMARY:
This study compared the effects of dairy products, including milk and yogurt, with different amounts of proteins on responses of appetite, glucose and insulin and on food intake at a meal served 120 minutes later in healthy adult male individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-30 years
* Body mass index: 20 and 24.9 kg/m2

Exclusion Criteria:

* Breakfast skippers,
* Smokers,
* Dieters,
* Individuals with lactose-intolerance or who are allergic to milk,
* Individuals with gastrointestinal problems and
* Individuals with diabetes or other metabolic diseases

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Food intake | 120 minutes after consumption of treatments
  Calories consumed at the test meal

SECONDARY OUTCOMES:
Glycemia | Pre-(0-120 min) and post-(120-260 min) meal periods
  Glycemic responses in the pre- and post-test meal periods

OTHER OUTCOMES:
Appetite | Pre-(0-120 min) and post-(120-260 min) meal periods
  Appetite scores in the pre- and post-test meal periods

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, Professor, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] El Khoury D, Brown P, Smith G, Berengut S, Panahi S, Kubant R, Anderson GH. Increasing the protein to carbohydrate ratio in yogurts consumed as a snack reduces post-consumption glycemia independent of insulin. Clin Nutr. 2014 Feb;33(1):29-38. doi: 10.1016/j.clnu.2013.03.010. Epub 2013 Mar 27. PMID 23591152